CLINICAL TRIAL: NCT07085546
Title: The Effects of Low-Flow Sevoflurane Anesthesia on Respiratory Mechanics, Gas Exchange, and Postoperative Pulmonary Function During One-Lung Ventilation: A Prospective Observational Study
Brief Title: Effects of Low-Flow Sevoflurane Anesthesia on Pulmonary Function During One-Lung Ventilation
Acronym: OLV-LOWSEVO
Status: Completed | Type: Observational
Sponsor: Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Eda Cennet Caferoğlu, Dr. - Department of Anesthesiology and Reanimation, Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital
Other Study IDs: 2025-05/56
Record Dates: First submitted 2025-07-12; First posted 2025-07-25 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: One-lung Ventilation (OLV); Low-flow Anesthesia; Thoracic Surgery; Respiratory Mechanics; Sevoflurane

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low-Flow Sevoflurane Group: Patients receiving low-flow sevoflurane anesthesia during one-lung ventilation
- Standard-Flow Sevoflurane Group: Patients receiving standard-flow sevoflurane anesthesia during one-lung ventilation

SUMMARY:
This prospective observational study aims to evaluate the effects of low-flow sevoflurane anesthesia on respiratory mechanics, gas exchange, and postoperative pulmonary function in patients undergoing one-lung ventilation (OLV) during thoracic surgery. The study will compare patients receiving low-flow sevoflurane anesthesia with those receiving standard-flow anesthesia, focusing on parameters such as lung compliance, arterial oxygen levels (PaO₂), and postoperative oxygen requirements.

Fifty patients scheduled for elective thoracic surgery with OLV will be included. Data will be collected intraoperatively and postoperatively, and standard anesthesia protocols will be followed according to the attending anesthesiologist's preference. The results are expected to provide new insights into the safety and efficacy of low-flow anesthesia protocols in thoracic surgery, potentially guiding future clinical practice to reduce postoperative pulmonary complications.

DETAILED DESCRIPTION:
One-lung ventilation (OLV) is a common technique used during thoracic surgery to optimize the surgical field and improve operative conditions. However, OLV is associated with potential complications such as hypoxemia, lung collapse, and inflammatory responses. The choice of anesthesia technique plays a critical role in minimizing these adverse effects.

Low-flow anesthesia (LFA), defined as the administration of inhalational anesthetics with a fresh gas flow rate of 1 L/min or less, offers several advantages, including reduced anesthetic consumption, better humidification of inspired gases, decreased heat loss, and more stable pulmonary gas exchange. Despite these benefits, concerns remain regarding the risk of hypoxemia and the need for careful monitoring of anesthesia depth during LFA.

This prospective, single-center, observational study will investigate the effects of low-flow sevoflurane anesthesia on respiratory mechanics, gas exchange, and postoperative pulmonary function in patients undergoing OLV for elective thoracic surgery. Patients will be allocated to either low-flow or standard-flow anesthesia groups based on routine clinical practice, without randomization. Standard anesthesia and ventilation protocols will be applied according to the attending anesthesiologist's preference.

Primary outcomes include intraoperative lung compliance, arterial oxygenation (PaO₂), and postoperative oxygen requirements. Secondary outcomes include the incidence of atelectasis, anesthetic gas consumption, and hemodynamic parameters. Data will be collected during both intraoperative and postoperative periods. The study aims to enroll 50 patients (25 per group), as determined by power analysis.

The findings of this study are expected to provide comprehensive data on the impact of low-flow sevoflurane anesthesia during OLV, particularly regarding respiratory mechanics and postoperative pulmonary function. These results may contribute to the development of safer and more effective anesthesia protocols for thoracic surgery patients.

ELIGIBILITY:
Inclusion Criteria:

Age between 18 and 75 years American Society of Anesthesiologists (ASA) physical status I-III Scheduled for elective video-assisted thoracoscopic surgery (VATS) or thoracotomy No acute respiratory failure

Exclusion Criteria:

Severe chronic obstructive pulmonary disease (COPD) or restrictive lung disease Body mass index (BMI) greater than 40 kg/m² Cardiac dysfunction with ejection fraction (EF) less than 40% Requirement for emergency thoracic surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 18 to 75 years who are scheduled for elective video-assisted thoracoscopic surgery (VATS) or thoracotomy under general anesthesia with one-lung ventilation at Dr. Abdurrahman Yurtaslan Oncology Training and Research Hospital. Eligible participants will have ASA physical status I-III and no acute respiratory failure.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2025-07-15 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Postoperative Oxygen Requirement | 24-hour postoperative period
Static Lung Compliance | Intraoperative period
  Static lung compliance (Cstat) will be calculated using the formula: Cstat = VT / (Pplateau - PEEP), where VT is tidal volume, Pplateau is plateau pressure, and PEEP is positive end-expiratory pressure
Arterial Oxygen Pressure (PaO₂) | Intraoperative period
  Arterial oxygen pressure (PaO₂) will be measured from arterial blood gas analysis during one-lung ventilation

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Abdurrahman Yurtaslan Oncology Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No